CLINICAL TRIAL: NCT03591055
Title: Frailty Assessment and Multimodal Treatment Strategies in the Elderly at Risk of Adverse Results and Functional Decline in the Community
Brief Title: Frailty Assessment and Treatment Strategies in the Elderly at Risk of Functional Decline in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI16/01683
Record Dates: First submitted 2018-06-22; First posted 2018-07-18 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Frail Elderly Syndrome
Keywords: Frail elderly; Clinical Trial
MeSH Terms: interventions — Medication Review; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group will be first derived to a nurse case manager for initial application of a comprehensive geriatric assessment. Then patient-centered interventions will be prescribed, according to the different target areas identified in the geriatric assessment. All participants in the intervention group will undergo a medication review and will also perform an aerobics exercise plan in the primary care centre, 60-minute session twice a week on non-consecutive days for 6 weeks (12 sessions of 60 minutes each) and memory workshops (10 sessions).
  Interventions: Other: CGA, medication review, exercise and cognitive stimulation
- Control group (No Intervention): Participants in the control group will receive the usual standard care and regular referrals.

INTERVENTIONS:
Other: CGA, medication review, exercise and cognitive stimulation — Comprehensive geriatric assessment. Patient-centered interventions according to the different target areas identified in the geriatric assessment. Medication review. Groupal Exercise plan and memory workshops.
  Arms: Intervention Group

SUMMARY:
This study aims to design a patient -centered program to prevent or delay frailty , functional decline and adverse events, and evaluates the effectiveness of the program with a randomized clinical trial.

DETAILED DESCRIPTION:
Objective: To design and evaluate the implementation and impact of a multimodal intervention focused on elderly patients living in the community in preventing or delaying frailty, functional decline and risk of institutionalization, hospitalization and death.

Design: Study in two phases: a qualitative study to develop the intervention and a randomized clinical trial with parallel arms and control group.

Intervention: Participants in the control group will receive the usual standard care and regular referrals. Patients in the intervention group will be first derived to a nurse case manager for initial application of a comprehensive geriatric assessment (CGA). Then patient-centered interventions will be prescribed, according to the different target areas identified in the geriatric assessment, along with medication review, aerobics exercise plan and memory workshops following the model adapted in Phase I.

After 3 and 18 months, measures of functional and cognitive performance, quality of life, frailty, adverse outcomes (institutionalization, hospitalization, death) and health care costs will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Positive screen in the accumulation of deficits electronic frailty index
* Positive screen with Gerontopole screening tool and/or RISC tool

Exclusion Criteria:

* Living in an institution
* Advanced conditions with short life expectancy
* Severe disability
* Severe Dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Short Physical Performance Battery (SPPB) at 3 and 18 months | 0, 3, 18 months
  The Short Physical Performance Battery (SPPB) is a standardised assessment tool of lower limb function, testing 3 dimensions: standing balance, walking speed, and chair stands. Each component is scored between 0-4, total score from 0 (poor performance) to 12 (best performance).
Change from Baseline in the Quick Mild Cognitive Impairment Screen (Qmci-S) at 3 and 18 months | 0, 3, 18 months
  The Quick Mild Cognitive Impairment (Qmci) screen is a multi-purpose, short cognitive screening instrument designed to differentiate between normal cognitive function, subjective cognitive disorders, mild cognitive impairment (MCI) and early dementia and to measure change over time.
Change from Baseline in Health Related Quality of Life (EuroQol 5D) at 3 and 18 months | 0, 3, 18 months
  EuroQol 5D EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.

SECONDARY OUTCOMES:
Change from Baseline in Functional Capacity at 3 and 18 months | 0, 3, 18 months
  Activities of daily living: Barthel Index and Lawton&Brody Index
Change from Baseline in the Risk Instrument for Screening in the Community (RISC) at 3 and 18 months | 0, 3, 18 months
  Risk Instrument for Screening in the Community is a validated short (2-5 min), global subjective assessment of risk created to identify patients' 1-year risk of three outcomes: institutionalization, hospitalization and death.
Change from Baseline in Clinical Frailty Scale (CFS) at 3 and 18 months | 0,3 18 months
  The clinical frailty scale is a 9 points measure of frailty based on clinical judgement.
Change from Baseline in the Gerontopole Frailty Screening Tool (GFST) at 3 and 18 months | 0,3,18 months
  Gerontopole Frailty Screening Tool is a questionnaire aimed to measure general signs and/or symptoms potentially indicating the presence of an underlying frailty. These questions largely mirror the criteria that are commonly used to operationalize the frailty status.

OTHER OUTCOMES:
Number of Participants Institutionalized during follow-up, at 18 months | 18 months
  Admission to long-term care {nursing home}
Number of Participants Hospitalized during follow-up, at 18 months | 18 months
  Hospitalization including prolonged admission or readmission
Number of Participants who die during follow-up, at 18 months | 18 months
  Death
Health care costs | 18 months
  Direct health care costs
Number of participants that comply with the programme schedules at 3 and 18 months | 3 months and 18 months
  Compliance with the programme: number of undergone interventions out of total prescribed interventions (including activities, referrals or prescriptions)
Number of participants (patients, caregivers and professionals) that are satisfied with the programme at 3 and 18 months | 3 months and 18 months
  Satisfaction with the programme, measured with an ad hoc questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCISCO Orfila Pernas, Principal Investigator — Institut Catala de Salut
Locations (1):
- IDIAP JGol, Barcelona, Spain